CLINICAL TRIAL: NCT02980432
Title: Verticality Perception - Modulatory Effect of a Rotating Optokinetic Stimulus on the Haptic Vertical in Healthy Human Subjects
Brief Title: Verticality Perception Assessed by the Haptic Vertical
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: shv_okn_study
Record Dates: First submitted 2016-11-16; First posted 2016-12-02 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Healthy
Keywords: vestibular; spatial orientation; vision; optokinetic
MeSH Terms: conditions — Orientation, Spatial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intervention arm (Experimental): all participants will be assigned to the same arm. Interventions applied include presenting a visual line or a rod with or without a moving (rotating) background while being in different whole-body roll positions. Participants will be asked to adjust the line or the rod along perceived direction of gravity.
  Interventions: Other: changes in whole-body roll position and visual/haptic stimuli presented

INTERVENTIONS:
Other: changes in whole-body roll position and visual/haptic stimuli presented — In different whole-body roll positions subjects will be presented a luminous line or a rod in combination with a moving or stationary background. Participants will be asked to align the line or the rod along perceived direction of gravity.

SUMMARY:
The investigators previously shown that a rotating optokinetic stimulus results in shifts of the subjective visual vertical in healthy human subjects. However, the origin of these shifts is still poorly understood. Both torsional displacement of the eyes and a shift in the internal estimate of direction of gravity have been proposed as potential explanations. Here the investigators use a vision-independent setup to differentiate between these two hypotheses, predicting no impact of a rotating stimulus on the subjective haptic vertical if torsion triggers the shift.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-65 years
* informed consent
* absence of exclusion criteria

Exclusion Criteria:

* peripheral-vestibular deficit
* disturbed consciousness
* history of sensory deficits
* visual field deficits
* other neurological or systemic disorder which can cause dementia or cognitive dysfunction
* intake of antidepressants, sedatives, or neuroleptics
* pregnancy, unless excluded by a negative pregnancy test
* known neck pain or status post neck trauma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-10; Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Adjustment errors of aligning a rod along perceived direction of gravity while an optokinetic stimulus is presented. | 60 minutes
  This outcome parameter focuses on the adjustment errors of the subjective haptic vertical while presenting a visual bias (i.e. an optokinetic rotatory stimulus).
Trial-to-trial variability of aligning a rod along perceived direction of gravity while an optokinetic stimulus is presented. | 60 minutes
  This outcome parameter focuses on the trial-to-trial variability of rod alignments along perceived direction of gravity when presenting a visual bias cue (i.e. an optokinetic rotatory stimulus).

SECONDARY OUTCOMES:
Comparison of adjustment errors between the subjective haptic vertical and the subjective visual vertical | 60 minutes
Comparison of adjustment errors of perceived vertical using the subjective haptic vertical with and without presenting an optokinetic stimulus | 60 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Dept. of Neurology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No